CLINICAL TRIAL: NCT02601833
Title: The Effectiveness of Silver Diamine Fluoride as a Treatment for Caries in Comparison to Traditional Restorative Techniques: A 12 Month Randomized Controlled Trial
Brief Title: Effectiveness of Silver Diamine Fluoride as a Treatment for Caries in Comparison to Traditional Restorative Techniques
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Mott Children's Health Center (Other)
Responsible Party: Principal Investigator, Margherita Fontana, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00097829
Record Dates: First submitted 2015-11-02; First posted 2015-11-10 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Caries
Keywords: Caries; Cavity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silver Diamine Fluoride (Experimental): This arm will receive Silver Diamine Fluoride applied to their carious lesion, in lieu of restoration placement, with the goal of arresting caries.
  Interventions: Device: Silver Diamine Fluoride
- Conventional Caries Management (Active Comparator): Restorative dental care according to American Academy of Pediatric Dentistry guidelines. This treatment typically includes administration of local anesthesia, placement of rubber dam, caries removal with rotary and hand instruments, and placement of a final restoration.
  Interventions: Procedure: Conventional Caries Management

INTERVENTIONS:
Device: Silver Diamine Fluoride — No caries removal will take place. The tooth will be dried and Silver Diamine Fluoride will be placed on the carious dentin until saturated. Excess will be blotted dry with a cotton pellet.
  Other Names: Silver Dental Arrest
  Arms: Silver Diamine Fluoride
Procedure: Conventional Caries Management — These children will receive restorative dental care in alignment with the American Academy of Pediatric Dentistry guidelines, within the confines of the Mott Children's Health Center clinic. This treatment typically includes administration of local anesthesia, placement of rubber dam, caries removal with rotary and hand instruments, and placement of a final restoration.
  Other Names: Filling; Restoration
  Arms: Conventional Caries Management

SUMMARY:
The purpose of this study is to compare standard fillings and silver diamine fluoride (SDF) for treatment of cavities in baby teeth. The investigators will compare the effectiveness of stopping the cavity, cost of the treatments and the opinions of the families and the dental providers.

DETAILED DESCRIPTION:
To determine the effectiveness of the application of silver diamine fluoride (SDF) in comparison to conventional restorative treatments in International Caries Detection and Assessment System criteria (ICDAS) 5 and 6, one and two surface carious lesions in primary molars which will be assessed based on major and minor failure criteria when followed for one year. Additionally, parents'/children's and providers' perceptions will be assessed as well as the cost of both regimens, to include both chair time spent and materials' costs.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one active (soft) cavitated carious lesions in the primary dentition, extending into dentin (ICDAS 5 or 6)
* The selected tooth must have a one or two surface lesion (more than 1/3 of the crown of the tooth must be remaining) and must allow for direct application of SDF
* Study teeth will not have any spontaneous or elicited pain due to caries, tooth mobility, or signs of pulpal infection
* Selected primary teeth must have an anticipated exfoliation date greater than 12 months away

Exclusion Criteria:

* Hereditary developmental defects such as Amelogenesis Imperfecta and Dentinogenesis Imperfecta
* Severe medical conditions that do not allow the child to be managed in the clinic
* Known allergy /sensitivity to dental materials being used, including SDF
* Inability of the child to cooperate for treatment, recall examinations, or periapical radiographs
* Wards of the State, for consenting reasons

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2016-01; Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margherita R Fontana, DDS, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan School of Dentistry, Ann Arbor, Michigan
  - Mott Children's Health Center, Flint, Michigan

REFERENCES:
- [Derived] Cleary J, Al-Hadidi R, Scully A, Yahn W, Zaid Z, Boynton JR, Eckert GJ, Yanca E, Fontana M. A 12-Month Randomized Clinical Trial of 38% SDF vs. Restorative Treatment. JDR Clin Trans Res. 2022 Apr;7(2):135-144. doi: 10.1177/23800844211072741. Epub 2022 Feb 4. PMID 35120408

RESULTS

PARTICIPANT FLOW:
Groups:
- Silver Diamine Fluoride: This arm will receive Silver Diamine Fluoride applied to their carious lesion, in lieu of restoration placement, with the goal of arresting caries. This is applied at baseline and at 6 Months.
  Silver Diamine Fluoride: No caries removal will take place. The tooth will be dried and Silver Diamine Fluoride will be placed on the carious dentin until saturated. Excess will be blotted dry with a cotton pellet.
- Conventional Caries Management: Restorative dental care according to American Academy of Pediatric Dentistry guidelines. This treatment typically includes administration of local anesthesia, placement of rubber dam, caries removal with rotary and hand instruments, and placement of a final restoration.
  Conventional Caries Management: These children will receive restorative dental care in alignment with the American Academy of Pediatric Dentistry guidelines, within the confines of the Mott Children's Health Center clinic and University of Michigan Pediatric Dental Clinic.
Period: Overall Study
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management
Started | 56 | 42
Completed | 40 | 29
Not Completed | 16 | 13

BASELINE CHARACTERISTICS:
Population: Treatment failures were assessed throughout the 12 month duration of the trial.
Groups:
- Silver Diamine Fluoride: This arm will receive Silver Diamine Fluoride applied to their carious lesion, at baseline and 6 months, in lieu of restoration placement, with the goal of arresting caries.
  Silver Diamine Fluoride: No caries removal will take place. The tooth will be dried and Silver Diamine Fluoride will be placed on the carious dentin until saturated. Excess will be blotted dry with a cotton pellet.
- Conventional Caries Management: Restorative dental care according to American Academy of Pediatric Dentistry guidelines. This treatment typically includes administration of local anesthesia, placement of rubber dam, caries removal with rotary and hand instruments, and placement of a final restoration.
  Conventional Caries Management: These children will receive restorative dental care in alignment with the American Academy of Pediatric Dentistry guidelines, within the confines of the Mott Children's Health Center clinic and the University of Michigan School of Dentistry.
- Total: Total of all reporting groups
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management | Total
Number analyzed (Participants) | 56 | 42 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 56 | 42 | 98
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.7 (1.9) | 4.8 (1.7) | 4.8 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 16 | 45
  Male | 27 | 26 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 51 | 40 | 91
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 22 | 54
  White | 14 | 16 | 30
  More than one race | 6 | 4 | 10
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 56 | 42 | 98
dmft [Mean (Standard Deviation); unit: dmft] — A measure of the number of baby teeth impacted by dental decay in a child patient. A larger number means more decay. The range is 0 to 20.
  dmft | 5.6 (3.7) | 7.2 (3.8) | 6.3 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Caries Arrest of Teeth in the SDF Group Measured by Change in Size
Description: Number of participants in the SDF arm that had an increase in lesion size at any point in the 12 months of the trial, as this is a treatment failure.
  Treatment failures were assessed throughout the 12 month duration of the trial, and children with treatment failures were then removed from the trial for further clinical treatment.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride
Number analyzed (Participants) | 56
Participants | 10

2. Primary Outcome: Caries Arrest of Teeth in the SDF Group Measured by Dentin Color (Yellow, Brown, Black)
Description: Color of the cavity at the end of the trial
Time Frame: 12 Months
Population: Only 39 of the 40 children who attended the 12 month visit in the SDF arm had cavities available for assessment. One child's tooth exfoliated (fell out) normally one week prior to the 12 month appointment.
  Please note dentin color cannot be assessed for the Conventional group as the dentin is no longer accessible following baseline treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride
Number analyzed (Participants) | 39
Participants
  Black | 37
  Brown | 0
  Yellow | 2

3. Primary Outcome: Caries Arrest of Teeth in the SDF Group Measured by Dentin Texture (Soft, Hard)
Description: Texture of the cavity's dentin of soft means the cavity is still an active infection. If the cavity is hard, the cavity is no longer an active infection (has been arrested).
  Please note dentin texture cannot be assessed for the Conventional group as the dentin is no longer accessible following baseline treatment.
Time Frame: 12 Months
Population: Only 39 of the 40 children who attended the 12 month visit in the SDF arm had cavities available for assessment. One child's tooth exfoliated (fell out) normally one week prior to the 12 month appointment.
  Dentin texture cannot be assessed for the Conventional group as the dentin is no longer accessible following baseline treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride
Number analyzed (Participants) | 39
Participants
  Soft Dentin | 10
  Hard Dentin | 29

4. Primary Outcome: Restoration Integrity for Teeth in Control Group (Secondary Caries, Lost Restoration, Restoration Needing Repair)
Description: Secondary caries, lost restorations, or restorations needing repair are treatment failures.
  Treatment failures were assessed throughout the 12 month duration of the trial, and children with treatment failures were removed from the trial for further clinical treatment.
Time Frame: 12 Months
Population: Please note restoration integrity cannot be assessed for the SDF group as this group does not receive a restoration.
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Caries Management
Number analyzed (Participants) | 42
Participants
  Missing restoration | 1
  Secondary caries and lesion progression | 1
  Intact restoration | 40

5. Primary Outcome: Signs of Pulpal Pathology (Lesion Reaching the Pulp Requiring Pulpular Treatment-pulpotomy and/or Pulpectomy-, Reversible Pulpitis, Irreversible Pulpitis, Abscess)
Description: Signs of pulpal pathology are treatment failures. Treatment failures were assessed throughout the 12 month duration of the trial, and children with treatment failures were removed from the trial for further clinical treatment.
Time Frame: 12 Months
Population: All children were assessed for signs of pulpal pathology throughout the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management
Number analyzed (Participants) | 56 | 42
Participants
  Reversible Pulpitis | 1 | 1
  Reversible Pulpitis and Later Periapical Infection | 2 | 0
  Periapical Infection | 2 | 0
  No Sign of Pulpal Pathology | 51 | 41

6. Secondary Outcome: Number of Providers Who Find Treatment With SDF More Favorable in Time for Treatment (More, Same, Less)
Description: Data collected at baseline only.
Time Frame: Baseline
Population: The 98 instances of treatment below were given by about 15 providers. The provider stated how much time each treatment instance took compared to the alternate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management
Number analyzed (Participants) | 56 | 42
Participants
  More time | 0 | 12
  Same amount of time | 1 | 27
  Less time | 55 | 3

7. Secondary Outcome: Number of Providers Who Find Treatment With SDF More Favorable in Ease of Treatment (Easier, Harder, Same Difficulty)
Time Frame: Baseline
Population: The 98 instances of treatment below were given by about 15 providers. The provider stated the ease of treatment for each treatment instance.
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management
Number analyzed (Participants) | 56 | 42
Participants
  Easier for the provider | 46 | 2
  The same level of difficulty for provider | 10 | 31
  Harder for the provider | 0 | 9

8. Secondary Outcome: Number of Providers Who Find Treatment With SDF More Favorable in Preference of Treatment Modality (More Preferable, no Preference, Less Preferable)
Time Frame: Baseline
Population: The 98 instances of treatment below were given by about 15 providers. The provider stated their treatment preference for each treatment instance.
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management
Number analyzed (Participants) | 56 | 42
Participants
  More preferable treatment for provider | 21 | 0
  No preference in treatment for provider | 35 | 41
  Less preferable treatment for provider | 0 | 1

9. Secondary Outcome: Parent Assessment of Appearance of Child's Teeth
Description: Parents were asked "Are you concerned with the appearance of your child's teeth?"
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management
Number analyzed (Participants) | 40 | 29
Participants
  No | 33 | 26
  Yes | 7 | 3

10. Secondary Outcome: Parent Assessment of Treatment Provided
Description: Parents were asked "If your child had another cavity, would you be willing to have that tooth treated with the same treatment option provided to your child in this study?"
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management
Number analyzed (Participants) | 40 | 29
Participants
  No | 7 | 3
  Yes | 33 | 26

11. Secondary Outcome: Child Assessment of Appearance of Teeth (Very Happy, Not Happy or Sad, Very Sad)
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management
Number analyzed (Participants) | 40 | 29
Participants
  Very Happy | 29 | 26
  Not Happy or Sad | 7 | 3
  Very Sad | 4 | 0

12. Secondary Outcome: Child Assessment of Experience During Dental Visit (Didn't Hurt, Hurt a Little, Hurt a Lot)
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management
Number analyzed (Participants) | 40 | 29
Participants
  Didn't Hurt at All | 27 | 25
  Hurt a Little | 10 | 4
  Hurt a Lot | 3 | 0

13. Secondary Outcome: Costs of Treatment (Dollars)
Description: Cost of one application of SDF and one 1-2 surface conventional restoration. Cost was calculated by taking the average Medicaid reimbursement across all U.S. states.
Time Frame: Baseline
Measure: Mean (Full Range); unit: Dollars
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management
Number analyzed (Participants) | 56 | 42
Dollars | 20.62 [2.71 to 98.50] | 79.68 [30.00 to 178.80]

14. Secondary Outcome: Time of Treatment Procedures (Duration of Time in Minutes)
Time Frame: Baseline
Measure: Mean (Full Range); unit: Time in Minutes
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management
Number analyzed (Participants) | 56 | 42
Time in Minutes | 5 [5 to 10] | 30 [17 to 40]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Patients were assessed clinically at baseline, 3, 6 and 12 months, and contacted at 1, 2, 4.5 and 9.5 months.
  Some categories below have 0 patients at risk of the AE due to the AE only pertaining to one of the treatment arms. The SDF group did not have a restoration, so it could not have a missing restoration or secondary caries on that restoration. The Conventional group's lesion was no longer accessible as it was covered with a restoration, and so the the lesion texture could not be assessed.
Arm/Group | Silver Diamine Fluoride | Conventional Caries Management
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/42
Other Adverse Events (participants affected / at risk) | 36/56 | 3/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Silver Diamine Fluoride (N=56) | Conventional Caries Management (N=42)
Radiographic signs of periapical infection (Infections and infestations) | 4 | 0 — Assessed at 12 months
Extraction (Infections and infestations) | 3 | 0 — Assessed at 12 months.
Active (soft) Lesion (Infections and infestations) | 25 | 0/0
Active (soft) Lesion with Progression (Infections and infestations) | 7 | 0/0
Hard (arrested) Lesion with Progression (Infections and infestations) | 3 | 0/0
Missing Restoration (Infections and infestations) | 0/0 | 1
Secondary caries and lesion progression (Infections and infestations) | 0/0 | 1
Reversible Pulpitis (Infections and infestations) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT02601833/Prot_SAP_000.pdf